CLINICAL TRIAL: NCT02640638
Title: Reducing Disparities in Birth Outcomes: a Randomized Controlled Trial of CenteringPregnancy
Brief Title: A RCT of CenteringPregnancy on Birth Outcomes
Acronym: CRADLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: Prisma Health-Upstate (Other); University of California, Los Angeles (Other); Georgia State University (Other)
Responsible Party: Principal Investigator, Moonseong Heo, Contact Principal Investigator, Clemson University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD082311 (NIH)
Record Dates: First submitted 2015-12-20; First posted 2015-12-29 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Pregnancy; Preterm Birth
Keywords: Racial disparities
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CenteringPregnancy group prenatal care (Experimental): Pregnant women who were randomized to receive CenteringPregnancy group prenatal care
  Interventions: Behavioral: CenteringPregnancy
- Traditional individual prenatal care (No Intervention): Pregnant women who were randomized to receive traditional individual prenatal care

INTERVENTIONS:
Behavioral: CenteringPregnancy — 8-12 pregnant women whose due dates are in the same month will receive ten 2-hour group prenatal care sessions according to the standard curriculum provided by the Centering Healthcare Institute.
  Arms: CenteringPregnancy group prenatal care

SUMMARY:
The purpose of this study is to evaluate whether CenteringPregnancy group prenatal care can improve preterm birth rate and other birth outcomes, maternal psychosocial and behavioral outcomes, and decrease the racial difference in selected birth outcomes among African American and White women, compared to individual prenatal care.

DETAILED DESCRIPTION:
This is a randomized controlled trial to compare biomedical, behavioral and psychosocial outcomes by race among pregnant women who participate in CenteringPregnancy group prenatal care, to women in the traditional individual prenatal care and to investigate whether improving women's stress, activation and engagement will explain the potential benefits of CenteringPregnancy on outcomes and health disparities. The trial will be conducted in a large prenatal care center in South Carolina. Eligible White and Black women will be recruited before 20 weeks of gestational age with low risk pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged between 14-45 years
2. Entry prenatal care before 20 6/7 weeks gestational age (defined as attendance at the intake screening visit). Patients must be randomized by 23 6/7 weeks gestational age.

Exclusion Criteria:

1. Medical complications of pregnancy that would preclude prenatal care provision by nurse practitioners or participation in group care

   * Pregestational diabetes,
   * Severe chronic hypertension requiring medication,
   * Morbid Obesity with BMI >49.99
   * Renal disease with baseline proteinuria >1g/24 hours
   * Any disease requiring chronic immunosuppression (SLE, solid organ transplant)
   * Active pulmonary tuberculosis
   * Sickle cell anemia
   * Human Immunodeficiency Virus Infection
   * Other medical conditions that would exclude women from group care at the discretion of the PI
2. Pregnancy complications that would preclude prenatal care provision by nurse practitioners or participation in group care

   * Multiple gestation
   * Lethal fetal anomalies
   * Other pregnancy complications that would exclude women from group care at the discretion of the PI
3. Social and behavioral complications of pregnancy which would preclude prenatal care provision by nurse practitioners or participation in group care

   * Current incarceration
   * Severe psychiatric illness

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2350 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Preterm birth | Measured at delivery
  Delivery before 37 weeks gestation

SECONDARY OUTCOMES:
Birth weight | Measured at delivery
  Infant weight (in grams) a birth
APGAR score | Measured at delivery
  Five criteria used to summarize the health of newborn children: Appearance, Pulse, Grimace, Activity, Respiration
Gestational weight gain | Measured at delivery
  Weight gained during pregnancy as compared to medical recommendation
Gestational diabetes incidence | Measured during pregnancy
  Diabetes (occurred during pregnancy (two steps: 50-g GLT (nonfasting) with PG measurement at 1 h (Step 1), at 24-28 wks in women not previously diagnosed with overt diabetes If PG at 1 h after load is ≥140 mg/dL (7.8 mmol/L), proceed to 100-g OGTT (Step 2), performed while patient is fasting GDM diagnosis made when two or more PG levels meet or exceed: Fasting: 95 mg/dL or 105 mg/dL (5.3/5.8)
  1. hr: 180 mg/dL or 190 mg/dL (10.0/10.6)
  2. hr: 155 mg/dL or 165 mg/dL (8.6/9.2)
  3. hr: 140 mg/dL or 145 mg/dL (7.8/8.0)
Gestational hypertension | Measured during pregnancy
  Hypertension (SBP/DBP: above 140/90 mm Hg) occurred during pregnancy according to medical chart
Patient activation measure | Measured at <20 week and 32-36 week of gestational age
  Based on self-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Moonseong Heo, PhD, Principal Investigator — Clemson University
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Georgia State University, Atlanta, Georgia
  - Clemson University, Clemson, South Carolina
  - Prisma Health, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be available publicly on the NICHD/DASH Data and Specimen Hub (https://dash.nichd.nih.gov/) in October 2026, five years after study completion. Prior to that time, researchers with a methodologically sound proposal can direct inquiries to amy.crockett@prismahealth.org to gain access to the study protocol, informed consent forms, deidentified data, data dictionaries and the analytic plan. Requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified study data will be available publicly on the NICHD/DASH Data and Specimen Hub (https://dash.nichd.nih.gov/) in October 2026, five years after study completion.
Access Criteria: Requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Hsieh CT, Zhang L, Britt J, Shodahl S, Crockett A, Chen L. Pregnancy Anxiety and Risk of Gestational Diabetes Mellitus Among a Diverse U.S. Cohort. J Womens Health (Larchmt). 2025 Jan;34(2):206-213. doi: 10.1089/jwh.2024.0453. Epub 2024 Oct 17. PMID 39419550
- [Derived] Doherty EA, Cartmell K, Griffin S, Heo M, Chen L, Britt JL, Crockett AH. Discrimination and Adverse Perinatal Health Outcomes: A Latent Class Analysis. Prev Chronic Dis. 2023 Nov 2;20:E96. doi: 10.5888/pcd20.230094. PMID 37917614
- [Derived] Keenan-Devlin L, Miller GE, Ernst LM, Freedman A, Smart B, Britt JL, Singh L, Crockett AH, Borders A. Inflammatory markers in serum and placenta in a randomized controlled trial of group prenatal care. Am J Obstet Gynecol MFM. 2023 Dec;5(12):101200. doi: 10.1016/j.ajogmf.2023.101200. Epub 2023 Oct 22. PMID 37875178
- [Derived] Chen Y, Crockett AH, Britt JL, Zhang L, Nianogo RA, Qian T, Nan B, Chen L. Group vs Individual Prenatal Care and Gestational Diabetes Outcomes: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2330763. doi: 10.1001/jamanetworkopen.2023.30763. PMID 37642966
- [Derived] Francis E, Johnstone MB, Convington-Kolb S, Witrick B, Griffin SF, Sun X, Crockett A, Chen L. Group Prenatal Care Attendance and Women's Characteristics Associated with Low Attendance: Results from Centering and Racial Disparities (CRADLE Study). Matern Child Health J. 2019 Oct;23(10):1371-1381. doi: 10.1007/s10995-019-02784-7. PMID 31236826
- [Derived] Chen L, Crockett AH, Covington-Kolb S, Heberlein E, Zhang L, Sun X. Centering and Racial Disparities (CRADLE study): rationale and design of a randomized controlled trial of centeringpregnancy and birth outcomes. BMC Pregnancy Childbirth. 2017 Apr 13;17(1):118. doi: 10.1186/s12884-017-1295-7. PMID 28403832